CLINICAL TRIAL: NCT06853392
Title: Evaluation of Socket Preservation Using Autogenous Dentin Graft With Collagen Sponge on Dental Implant Stability
Brief Title: Socket Preservation Using Dentin Graft Autogenous Dentin Graft With Collagen Sponge on Dental Implant Stability AUTOGENOUS TOOTH GRAFT WITH COLLAGEN SPONGE ON DENTAL IMPLANT STABILITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Collaborators: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Amira Ali El said, teaching assistant, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P-ME-23-02
Record Dates: First submitted 2025-02-27; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Bone Loss; Bone Remodeling Disorder; Bone Resorption
Keywords: socket preservation; alveolar ridge defect; Dentin graft; Demineralized freeze dried allograft
MeSH Terms: conditions — Bone Diseases, Metabolic; Bone Resorption

STUDY DESIGN:
Intervention Model Description: test group :socket preservation by dentin graft covered with collagen sponge control group :socket preservation by demineralized freeze dried allograft covered by collagen sponge
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- demineralized freeze dried allograft (Active Comparator): demineralized freeze dried allograft with collagen sponge
  Interventions: Combination Product: Demineralized freeze dried allograft with collagen sponge
- autogenous dentin graft (Active Comparator): Autogenous dentin graft with collagen sponge
  Interventions: Combination Product: autogenous dentin graft with collagen sponge

INTERVENTIONS:
Combination Product: Demineralized freeze dried allograft with collagen sponge — Demineralized freeze dried allograft,filling 2/3 of the socket covered with collagen sponge ,six months, one time
  Other Names: DFDBA
  Arms: demineralized freeze dried allograft
Combination Product: autogenous dentin graft with collagen sponge — autogenous mineralized dentin graft, filling 2/3 of the socket covered with collagen sponge , six months, one time
  Other Names: ADG
  Arms: autogenous dentin graft

SUMMARY:
The present study was performed to evaluate socket preservation using collagen sponge with autogenous dentin graft versus collagen sponge with de-mineralised freez-dried bone graft on dental implant stability

DETAILED DESCRIPTION:
in our study we made socket preservation using two different grafts in two groups.

before grafting we took CBCT

we used autogenous dentin graft covered by collagen sponge in one group and demineralized freeze - dried allograft covered with collagen sponge in the other group.

after 6 months we Took another CBCT to assist the dimensional changes and bone density in the alveolar socket after grafting We inserted the implant and during insertion we took a core biopsy with trephine bur with external diameter 3 mm for histological analysis.

After implant insertion we assisted the stability using RFA.

ELIGIBILITY:
Inclusion Criteria:

* Patients are free from any systemic diseases.
* Patients with good oral hygiene.
* Age range from 25-50 years.
* Adequate inter arch space .

Exclusion Criteria:

* Medications that may affect bone turnover, and bone metabolic diseases.
* Smoker patients and alcoholics.
* Patients with parafunctional habits.
* Patients with active acute infection related to tooth of interest.
* Patients with a lack of compliance, and serious mental or psychological problems.
* Pregnant females.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
change in radiographic Socket dimensions from base line to 6 months | 6 months following the end of treatment
  CBCT measuring socket dimensions
change in bone density from base line to 6 months | 6 months following the end of treatment
  CBCT measuring bone density within the socket

SECONDARY OUTCOMES:
new bone formation | after six months at the time of implant placement
  Histological analysis for new bone formation by masson trichrome
implant stability | after six months at the time of implant placement
  measuring primary Implant Stability by resonance frequency analysis

CONTACTS AND LOCATIONS:
Locations (1):
- AL Azhar university for girls, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided